CLINICAL TRIAL: NCT04008056
Title: Impact of Patient Reported Outcomes for Pre-chemotherapy Medical Decision in Day Patients With Digestive Cancer
Acronym: PRO Link
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NIMAO/2017-03/MF-01
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2021-08

CONDITIONS: Digestive Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing chemotherapy (Experimental)
  Interventions: Other: Patient Reported Outcome questionnaire

INTERVENTIONS:
Other: Patient Reported Outcome questionnaire — 34 question form to assess patient symptoms

SUMMARY:
The investigators hypothesize that an early assessment of the clinical toxicity of the patient is possible via patient reported outcomes and that this information provides at least the same information level as the clinical examination of the patient made by the doctor. The early decision to prepare chemotherapy medications based on the indirect early collection of clinical information from the patient via a patient reported outcome should help minimize the number of chemotherapy medications destroyed.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient is undergoing at least their second chemotherapy regime (outside weekly scheme or protocol with cisplatin requiring hospitalization) for a digestive tumor
* Patient has a Smartphone or access to the internet (via tablet or computer)
* The patient is under consultation as a day patient in the Oncology Department of Nimes hosptial

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant, parturient or breastfeeding
* Patient has already participated in the study
* Patient undergoing first chemotherapy regime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-11-16 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Authorization for preparation of chemotherapy based on clinical information (decision 2) | Day 1
  Yes/no
Authorization for preparation of chemotherapy based on patient reported outcome (decision 3) | Day 1
  Yes/no

SECONDARY OUTCOMES:
Cost of unused pouches of prepared chemotherapy according to decisions | Day 1
  Euros
Authorization for preparation of chemotherapy based on biological results (decision 1) | Day 0
  Yes/no
Patient satisfaction with the patient reported outcome questionnaire | Before starting chemotherapy (Up to 72 hours prior to treatment starting)
  System Usability Scale (SUS); score between 0-100 where the higher the score, the more satisfied the patient is.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Favier, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France